# Cognitive Stimulation Therapy for Residents With Dementia in Skilled Nursing Facilities: A Quasi-Experimental Study

NCT06978972

June 26, 2025

### PARTICIPANT CONSENT TO PARTICIPATE IN RESEARCH

**STUDY TITLE:** Cognitive Stimulation Therapy for Residents With Dementia in Long-Term Facilities: A Quasi-Experimental Study

NAME OF STUDENT RESEARCHER(s): Michael Agee, OTS; Abigail Halsey, OTS, MA; Jenna Range, OTS; Zoe Webb, OTS

FACULTY ADVISORY: Terrance Anderson, OTD, MS, OTR/L

TELEPHONE Number/Email Address: 937-781-6940/halseya2@mymail.nku.edu

Funding Organization: Northern Kentucky University

#### KEY INFORMATION

<u>Study Purpose:</u> This study led by occupational therapy students will use Cognitive Stimulation Therapy (CST) at your facility. The goal is to find out if CST increases your memory, thinking skills, ability to perform daily activities, and socialization.

<u>Major Requirements of the Study:</u> To participate in this student-led project, you must be diagnosed with mild to moderate dementia. You should also be older than 18 years old, and speak and understand English well.

Significant Risks: The activities in this study are considered safe and low-risk for injury.

<u>Potential Benefits:</u> By participating, you may experience an increase in socialization, thinking skills like memory, and ability to perform daily tasks.

<u>Duration of Participation:</u> 2 sessions per week (45-60 minutes per session) for 7 weeks for a total of 14 sessions.

#### Introduction

You are invited to join in a research study by Michael Agee, Abigail Halsey, Jenna Range, Zoe Webb, and Dr. Terrance Anderson from the Doctor of Occupational Therapy Program at Northern Kentucky University. Please read this form before joining and ask questions if you do not understand anything.

## Why are we doing this research?

In this research study, we want to learn more about cognitive stimulation therapy (CST) and its effects on people with mild-to-moderate dementia. We are looking at how CST affects the ability to participate in activities, engage with others, and improve thinking skills. There is limited research on occupational therapists (OTs) using CST for individuals with dementia in nursing homes in the United States, so we want to learn more. We aim to improve care, cognition, independence, and quality of life for this population.

We are asking you and other people ages 18 years and older with a diagnosis of mild-to-moderate dementia to be in our research. To join, you need to live in a nursing home, participate in recreational activities, understand and speak English well, have good vision, hearing, and speech, and tolerate at least one hour of therapy.

WHO SHOULD BE IN THE RESEARCH?

Individuals who are 18 years or older with diagnosed mild-to-moderate dementia can join the study. They must live in a nursing home, engage in at least 45 minutes of recreational or social activities each week, and score in the mid-range on the Alzheimer's Disease Assessment Scale–Cognitive Subscale (ADAS-Cog). Additionally, they should speak English well and have good vision, hearing, and speech to participate in group activities. Participants and their POA (if applicable) must also provide informed consent by signing this form to be included in the study.

## WHO SHOULD NOT BE IN THE RESEARCH?

You cannot join this study if you: are 17 years of age or younger; are not receiving maintenance or recreational services; have communication barriers; do not speak English as a first or second language, do not have a dementia diagnosis; have a severe case of dementia, receive hospice care; score in the high range on the ADAS-Cog; had CST treatment before; have a history of brain injury or learning disability; and are participating in other research that may influence outcomes that are being tested. The criteria above are to ensure the right participants are in the study and to keep the results accurate.

## WHAT WILL YOU DO IN THE RESEARCH?

If you decide to take part in this study, here is what will happen: You will participate in a 7-week long group program, which will be performed at your facility by trained students under the supervision of an occupational therapist. Each week, the students will choose activities that evidence has shown to improve cognition or delay memory loss. Before the program starts, researchers will test your level of thinking skills and memory, noting any areas that may need improvement. In each session, you will participate in group activities for approximately 45 to 60 minutes. The sessions will consist of a 10-minute introduction followed by 25 minutes of activities and a 10-minute summary. After 7 weeks, researchers will check your thinking skills and note any changes from the first test. Researchers want to see if CST impacts the level of cognition. Based on the study, we will find out if CST helps people with dementia reduce cognitive impairment and/or slow down the effects of dementia.

## How long will you be in this research?

Participation will take approximately 2 sessions per week (45-60 minutes per session), for 7 weeks, for a total of 14 sessions.

## WHAT OTHER CHOICES ARE THERE?

Joining this study is up to you. At any point during the seven weeks, you can change your mind and quit the study group without punishment. You can say no to participating in treatment sessions for any reason. During any session, you can change your mind, leave the session, and/or quit the study altogether. We want you to join in during the sessions and will try to make activities fun, but you are allowed to skip any group activities.

You can also skip any questions you do not wish to answer. Whatever you decide will not punish you or result in loss of benefits or services to which you deserve.

# WHAT ARE THE BAD THINGS THAT CAN HAPPEN FROM THIS RESEARCH?

Based on past research, there have been no reported harmful side effects from participating in CST. This means that there is a low risk of harm from joining this study. If something bad were to happen, then we will follow HIPPA Law and your facility's rules. We will also report the incident or injury to the faculty advisor.

There is a small chance that your personal information could be accidentally shared; however, the researchers are taking steps to protect your data.

WHAT ARE THE GOOD THINGS THAT CAN HAPPEN FROM THIS RESEARCH?

Cognitive Stimulation Therapy may improve cognition and memory, quality of life, mental health, social interactions, and overall daily functioning. By joining this study, you may receive this treatment, which may reduce symptoms of dementia and depression, delay cognitive decline, and improve your quality of life. CST is a proven holistic treatment that does not require medicine. You can use CST if you want a natural way to manage your condition. CST can be used in addition to your medicine to help prevent or delay various symptoms.

This research may further the understanding of dementia and identify a treatment approach that works for dementia.

## How will information about you be kept private?

Confidentiality cannot be guaranteed: Because of the kind of data, we cannot promise that your data will stay private. It may be possible that others will know what you have reported. We will make every effort to ensure that your information remains private, but we cannot guarantee total confidentiality. Your name and identity will not be in any reports for publication. However, it may be possible for someone to recognize your story/situation/response. We will ask all group members to keep the information they hear in this group private, but we cannot guarantee that everyone will do so.

We will take the following measures to protect your information: files with names will be encrypted and moved to a secure system, and your name will be changed to a code. Only the students of the research team and faculty advisor will have access to your information through a password-protected flash drive. Your name will not be included on data collection sheets, only the ID. Documents containing your name will be stored in the faculty advisor's office and on a flash drive that is password-protected, protecting your privacy. After the completion of the study, data will be kept for six years. Paper documents will be shredded and devices where data is stored will be erased afterwards.

We would like your permission to keep your data for future research studies related to this one. If you agree, then your data will be stored in the faculty advisor's office on a password-protected flash drive.

# WILL YOU BE PAID TO BE IN THIS RESEARCH STUDY?

You will not be paid for participating in this study.

# WILL WE SHARE THE RESEARCH RESULTS WITH YOU?

The information we learn in this study could be important for your health and well-being. You will get a paper copy of the finalized research. You may need to talk to professionals to understand the results.

## WHAT HAPPENS IF YOU ARE INJURED FROM BEING IN THIS RESEARCH?

The activities we will do at your facility are safe and low-risk for harm. If you or someone else gets injured, then the rules of the facility will be followed.

## MANDATED REPORTING

We are mandated reporters. This means that if we learn or think that you are being abused or neglected, we must tell the authorities.

## WHO DO YOU CALL IF YOU HAVE QUESTIONS OR PROBLEMS?

If you have questions about this research, please contact the primary communication coordinator, Michael Agee, OTS, at: <a href="mailto:ageem2@nku.edu">ageem2@nku.edu</a>. You may also contact the faculty member supervising this work: Terrance Anderson, OTD, MS, OTR/L, at <a href="mailto:andersont13@nku.edu">andersont13@nku.edu</a>.

If you have any questions regarding your rights as a research participant, please contact the Chair of NKU's IRB, Andrea Lambert South, Ph.D., 859-572-6615 or <a href="mailto:irbchair@nku.edu">irbchair@nku.edu</a>.

#### **SIGNATURES**

| Signing this document means that you understand the information given to you in the voluntarily agree to participate in the research described above. | nis form and that you |
|---|---|
| <u>Participant</u> | |
| Printed Name of Research Participant | |
| Signature of Research Participant Indicating Consent | Date |
| Study Staff | |
| Signature of Individual Obtaining Consent Please sign both consent forms, keeping one for yourself | Date |